CLINICAL TRIAL: NCT01320202
Title: A Randomized, Placebo-Controlled, Phase III Study of Dialysate Containing Soluble Ferric Pyrophosphate (SFP) in Chronic Kidney Disease Patients Receiving Hemodialysis: The Continuous Replacement Using Iron Soluble Equivalents (CRUISE 1) Study
Brief Title: Continuous Soluble Ferric Pyrophosphate (SFP) Iron Delivery Via Dialysate in Hemodialysis Patients
Acronym: CRUISE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMTI-SFP-4
Record Dates: First submitted 2011-03-20; First posted 2011-03-22 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: End Stage Renal Disease; Hemodialysis; SFP; Hemodialysis-dependent chronic renal failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soluble Ferric Pyrophosphate (SFP) in dialysate (Active Comparator): 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Interventions: Drug: Soluble Ferric Pyrophosphate (SFP)
- Standard Dialysate (Placebo Comparator): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Interventions: Device: Standard dialysate

INTERVENTIONS:
Drug: Soluble Ferric Pyrophosphate (SFP) — Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 18 months.
  Arms: Soluble Ferric Pyrophosphate (SFP) in dialysate
Device: Standard dialysate — Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week.
  Arms: Standard Dialysate

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Soluble Ferric Pyrophosphate (SFP) dialysate solution in maintaining iron delivery for erythropoiesis in anemic adult patients with chronic kidney disease (CKD) receiving hemodialysis. Efficacy will be measured primarily by the change from baseline in hemoglobin (Hgb).

DETAILED DESCRIPTION:
Screening: 2-3 weeks prior to enrollment in Stage 1.

Stage 1 (Run-In): 1-4 weeks depending on qualification for Stage 2.

Stage 2 (Randomized Blinded Treatment): 12 months unless withdrawn prematurely.

Stage 3 (Open-Label Treatment): The duration of Stage 2 plus Stage 3 is intended to be 18 months regardless of treatment assignment in Stage 2.

ELIGIBILITY:
Stage 1:

Main Inclusion Criteria:

* Adult subject ≥ 18 years of age undergoing chronic hemodialysis three or four times per week for chronic kidney disease (CKD) for at least 4 months, and expected to remain on hemodialysis three to four times weekly and be able to complete the duration of the study.
* Received IV iron therapy between 6 months and 2 weeks prior to enrollment in order to replace iron losses resulting from hemodialysis procedure.
* Mean Screening Hgb ≥ 9.5 to ≤ 11.5 grams per deciliter (g/dL).
* Mean Screening Transferrin Saturation (TSAT) ≥ 15% to ≤ 40%.
* Mean Screening serum ferritin ≥ 200 to ≤ 800 micrograms per liter (µg/L).
* If being administered epoetin, darbepoetin, or CERA, epoetin dose ≤ 45,000 Units (U)/week, darbepoetin dose ≤ 200 micrograms (µg)/week, or CERA dose ≤ 400 micrograms (µg)/month during the four weeks prior to enrollment.

Main Exclusion Criteria:

* Patient has living kidney donor identified or living-donor kidney transplant scheduled. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
* Vascular access for dialysis with femoral catheter or non-tunneled catheter.
* Received a total of > 800 milligrams (mg) IV iron during the 8 weeks prior to enrollment
* If being administered an ESA, route of administration change or ESA dose change > 35% (i.e., [max - min dose]/max dose > 0.35) over the 2 weeks prior to screening.
* Serum albumin < 3.0 grams per deciliter (g/dL) any time over the 8 weeks prior to enrollment.
* Red Blood Cell (RBC) or whole blood transfusion within 12 weeks prior to enrollment.

Stage 2:

Main Inclusion Criteria:

* Patient currently enrolled in the Stage 1 run-in period of study.
* Undergoing chronic hemodialysis three or four times per week for chronic kidney disease (CKD), and expected to remain on hemodialysis three to four times weekly and be able to complete duration of the study.
* Mean Hgb ≥ 9.5 to ≤ 11.5 g/dL over the three most recent consecutive every-week measurements prior to randomization.
* Stable Hgb defined as ≤ 1.0 g/dL difference between the maximum and minimum Hgb values over the 3 weeks immediately prior to randomization.
* Mean TSAT ≥ 15% to ≤ 40% over the two most recent consecutive every-other-week measurements prior to randomization.
* Mean serum ferritin ≥ 200 to ≤ 800 µg/L over the two most recent consecutive every-other-week measurements prior to randomization.
* If being administered epoetin, darbepoetin, or CERA, epoetin dose ≤ 45,000 U/week, darbepoetin dose ≤ 200 µg/week, or CERA dose ≤ 400 µg/month during the four weeks prior to randomization.

Main Exclusion Criteria:

* Patient has living kidney donor identified or living-donor kidney transplant scheduled. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
* Vascular access for dialysis with femoral catheter or non-tunneled catheter.
* Received any amount of IV iron during the 4 weeks prior to randomization.
* If being administered an (Erythropoietin Stimulating Agent) ESA, change in dose over the 6 weeks immediately prior to randomization.
* Serum albumin < 3.0 g/dL any time over the 8 weeks prior to randomization.
* RBC or whole blood transfusion during Stage 1.

Stage 3:

Main Inclusion Criteria:

* Patient randomized in Stage 2 who has completed the full duration of Stage 2 and less than 4 weeks have elapsed since completion of Stage 2, OR
* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for protocol-defined Protocol-Mandated Change in Anemia Management and less than 4 weeks have elapsed since withdrawal from Stage 2, OR
* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for Hgb >11.5 g/dL over ≥ 1 week confirmed by ≥ 2 consecutive measurements AND an associated increase in Hgb by ≥ 1 g/dL over 4 weeks.

Main Exclusion Criteria:

* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for any reason other than as noted in inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-03; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Pratt, MD, Study Director — Rockwell Medical
Locations (44):
- United States (42):
  - Bakersfield, California
  - Investigative Site, Chula Vista, California
  - Cudahy, California
  - Downey, California
  - Encino, California
  - Los Angeles, California
  - National City, California
  - Northridge, California
  - Ontario, California
  - Panorama City, California
  - Riverside, California
  - San Dimas, California
  - Simi Valley, California
  - West Covina, California
  - Yuba City, California
  - Investigative Site, Waterbury, Connecticut
  - Waterbury, Connecticut
  - Coral Springs, Florida
  - Miami, Florida
  - Investigative Site, Augusta, Georgia
  - Chicago, Illinois
  - Michigan City, Indiana
  - Detroit, Michigan
  - Las Vegas, Nevada
  - Investigative Site, Mineola, New York
  - Investigative Site, Ridgewood, New York
  - Rosedale, New York
  - Yonkers, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - Arlington, Texas
  - Fort Worth, Texas
  - Investigative Site, Houston, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Shorewood, Wisconsin
- Puerto Rico (2):
  - Caguas
  - Carolina

REFERENCES:
- [Derived] Fishbane SN, Singh AK, Cournoyer SH, Jindal KK, Fanti P, Guss CD, Lin VH, Pratt RD, Gupta A. Ferric pyrophosphate citrate (Triferic) administration via the dialysate maintains hemoglobin and iron balance in chronic hemodialysis patients. Nephrol Dial Transplant. 2015 Dec;30(12):2019-26. doi: 10.1093/ndt/gfv277. Epub 2015 Jul 13. PMID 26175145

RESULTS

PARTICIPANT FLOW:
Groups:
- Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 48 weeks.
- Standard Dialysate: 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 48 weeks.
Period: Overall Study
Arm/Group | Soluble Ferric Pyrophosphate (SFP) in Dialysate | Standard Dialysate
Started | 152 | 153
Comp 48 Wks in St 2 | 27 | 27
Comp St 2 Due to ESA/IV Iron Needs | 69 | 82
Enrolled in St 3 | 98 | 109
Completed St 3 | 79 | 82
Completed | 96 | 109
Not Completed | 56 | 44
Not completed — Adverse Event | 5 | 5
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 10 | 3
Not completed — non-protocol change to ESA or IV iron | 17 | 20
Not completed — kidney transplant | 1 | 2
Not completed — blood transfusion | 1 | 7
Not completed — moved/changed dialysis | 5 | 2
Not completed — sponsor request | 2 | 0
Not completed — ineligible | 3 | 0
Not completed — regained renal function | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: all randomized subjects, regardless of whether they received any investigational product.
Groups:
- Standard Dialysate: 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 18 months.
- Total: Total of all reporting groups
Arm/Group | Soluble Ferric Pyrophosphate (SFP) in Dialysate | Standard Dialysate | Total
Number analyzed (Participants) | 152 | 153 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (12.56) | 59.9 (13.01) | 58.3 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 98
  Male | 102 | 105 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 65 | 139
  Not Hispanic or Latino | 78 | 88 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 12 | 18
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 50 | 48 | 98
  White | 84 | 84 | 168
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 145 | 143 | 288
  Puerto Rico | 7 | 10 | 17
post-dialysis body weight [Mean (Standard Deviation); unit: kilograms] | 84.08 (23.264) | 83.15 (22.166) | 83.61 (22.685)
height [Mean (Standard Deviation); unit: centimeters] | 168.48 (10.197) | 169.17 (9.350) | 168.82 (9.771)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hemoglobin at End-of-Treatment: Least-Squares Mean
Description: Mean change from baseline Hgb (the average of the three most recent Hgb values preceding randomization) assessments during the last one-sixth of the treatment period for patients who prematurely withdraw from study treatment, but will include a minimum of at least the last two Hgb values. Value is expressed as least-squares mean with standard error.
Time Frame: Hgb measured weekly; up to 48 weeks from the date of randomization
Population: modified intent-to-treat populations: all randomized subjects who received at least one dose of study medication and had at least one post-dose hemoglobin measurement obtained.
Measure: Least Squares Mean (Standard Error); unit: grams per liter
Groups:
- Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 48 weeks.
- Stage 2 Placebo (Standard Dialysate): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 48 weeks.
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
grams per liter | 0.6 (1.15) | -3.0 (1.14)
Statistical Analysis 1: Comparison: Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate vs Stage 2 Placebo (Standard Dialysate); Test type: Superiority or Other; p = 0.011, ANCOVA — LS Mean (SE) and p-value are from ANCOVA model with baseline Hgb as covariate. Model also includes indicator variable for baseline ESA dose stratum; Difference in LS Means between SFP & PBO = 3.6, Standard Error of Mean 1.40

2. Secondary Outcome: Mean Change in Serum Iron From Pre-dialysis to Post-dialysis.
Description: The mean difference between the pre-dialysis and post-dialysis serum iron was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from the date of randomization
Population: modified intent-to-treat population: all randomized subjects who received at least one dose of study drug and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
micromoles per liter
  mean pre-dialysis serum iron | 12.1 (4.15) | 10.8 (3.04)
  mean post-dialysis serum iron | 29.6 (8.64) | 11.5 (3.91)
  serum iron change from pre- to post-dialysis | 17.5 (8.70) | 0.6 (3.08)

3. Secondary Outcome: Mean Change in TSAT (Transferrin) From Pre-dialysis to Post-dialysis.
Description: The mean difference between the pre-dialysis and post-dialysis TSAT (transferrin) was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from the date of randomization
Population: modified intent-to treat: all randomized subjects who had at least one dose of study drug and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
percent
  mean pre-dialysis TSAT(transferrin) | 24.9 (6.86) | 22.4 (5.97)
  mean post-dialysis TSAT(transferrin) | 57.9 (15.94) | 22.2 (7.80)
  pre- to post-dialysis change in TSAT | 32.7 (15.83) | -0.4 (6.86)

4. Secondary Outcome: Mean Change in Unsaturated Iron Binding Capacity (UIBC) From Pre- to Post-dialysis.
Description: The mean difference between the pre-dialysis and post-dialysis unsaturated iron binding capacity (UIBC) was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from the date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study drug and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
micromole per liter
  mean pre-dialysis UIBC | 31.49 (6.797) | 32.27 (6.580)
  mean post-dialysis UIBC | 19.48 (7.911) | 34.51 (7.208)
  pre- to post-dialysis change in UIBC | -11.86 (6.604) | 2.38 (3.253)

5. Secondary Outcome: Red Blood Cell or Whole Blood Transfusion: Number of Patients Receiving Transfusion
Description: The number of patients requiring red blood cell or whole blood transfusion while in the randomized treatment stage (Stage 2). Patients remained in Stage 2 until they met protocol-defined criteria for Stage 2 completion or until they had participated in Stage 2 for 48 weeks (whichever came sooner). If a patient was transfused, they were withdrawn from Stage 2.
Time Frame: up to 48 weeks from the date of randomization
Population: Intent-to-Treat (ITT): all patients randomized are included.
Measure: Number; unit: participants
Groups:
- Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 48 weeks in Stage 2.
- Stage 2 Placebo (Standard Dialysate): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 48 weeks in Stage 2.
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 152 | 153
participants | 3 | 11

6. Secondary Outcome: Red Blood Cell or Whole Blood Transfusion: Number of Units Transfused
Description: The total number of units of red blood cells or whole blood that were received by patients while in the randomized treatment stage (Stage 2). This number is the total number of units received across all randomized patients in each treatment group (it is not the average number of units received per patient). Patients remained in Stage 2 until they met protocol-defined criteria for Stage 2 completion or until they had participated in Stage 2 for 48 weeks (whichever came sooner). If a patient was transfused, they were withdrawn from Stage 2.
Time Frame: up to 48 weeks from the date of randomization
Population: Intent-to-Treat (ITT): all patients randomized are included.
Measure: Number; unit: units of red blood cells or whole blood
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 152 | 153
units of red blood cells or whole blood | 5 | 19

7. Secondary Outcome: Percentage of Change From Baseline to End-of-Treatment (EoT) for: Reticulocyte Hemoglobin Content (CHr), Ferritin, and Pre-Dialysis Serum Iron Panel
Description: A comparison of the lab values at the end-of-treatment (EoT) to baseline was performed, and the percentage of change from baseline was calculated for the following lab parameters: reticulocyte hemoglobin content (CHr), Ferritin, pre-dialysis unbound iron-binding capacity (UIBC), pre-dialysis serum iron, pre-dialysis transferrin, pre-dialysis total iron-binding capacity TIBC), and transferrin saturation (TSAT).
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
percentage of change
  CHr: % of change from baseline | -0.64 (3.800) | -2.73 (4.289)
  Ferritin: % of change from baseline | -14.8 (27.68) | -28.5 (34.35)
  Pre-dialysis UIBC: % of change from baseline | 8.36 (53.186) | 7.62 (14.818)
  Pre-dialysis serum iron: % of change from baseline | 4.644 (53.1728) | -4.628 (29.0307)
  Pre-dialysis transferrin: % change from baseline | 1.718 (8.5133) | 2.633 (9.7691)
  Pre-dialysis TIBC: % of change from baseline | 1.80 (9.255) | 2.88 (10.253)
  Pre-dialysis TSAT: % of change from baseline | 1.8 (44.99) | -7.8 (26.42)

8. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Unsaturated Iron-Binding Capacity (UIBC), Serum Iron, and Total Iron-Binding Capacity (TIBC)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Unsaturated Iron-Binding Capacity (UIBC), Pre-Dialysis Serum Iron, and Pre-Dialysis Total Iron-Binding Capacity (TIBC) will be quantified.
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
micromoles per liter
  Baseline UIBC | 30.91 (6.784) | 30.77 (6.452)
  EoT UIBC | 32.76 (13.734) | 33.03 (7.527)
  UIBC: Change from Baseline to EoT | 1.93 (13.265) | 2.14 (4.447)
  Baseline Serum Iron | 11.976 (3.9192) | 11.443 (3.9198)
  EoT Serum Iron | 11.911 (4.5412) | 10.389 (3.4941)
  Serum Iron: Change from Baseline to EoT | -0.196 (4.7462) | -1.051 (3.6562)
  Baseline TIBC | 42.88 (7.458) | 42.22 (7.380)
  EoT TIBC | 43.59 (8.140) | 43.40 (7.964)
  TIBC: Change from Baseline to EoT | 0.65 (4.051) | 1.08 (4.296)

9. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Reticulocyte Hemoglobin Content (CHr)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Reticulocyte Hemoglobin Content (CHr) will be quantified.
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
picograms
  Baseline CHr | 32.37 (1.985) | 32.57 (1.953)
  EoT CHr | 32.12 (2.016) | 31.64 (2.019)
  CHr: Change from Baseline to EoT | -0.23 (1.203) | -0.91 (1.413)

10. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Ferritin
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Ferritin will be quantified.
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
micrograms per liter
  Baseline Ferritin | 509.6 (194.16) | 511.3 (209.68)
  EoT Ferritin | 440.7 (216.41) | 366.9 (224.01)
  Ferritin: Change from Baseline to EoT | -72.3 (133.40) | -143.1 (188.28)

11. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin will be quantified.
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
grams per liter
  Baseline Pre-Dialysis Transferrin | 1.928 (0.3427) | 1.908 (0.3475)
  EoT Pre-Dialysis Transferrin | 1.958 (0.3767) | 1.957 (0.3731)
  Pre-Dialysis Ferritin: Change from Baseline to EoT | 0.029 (0.1695) | 0.044 (0.1883)

12. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin Saturation (TSAT)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin Saturation (TSAT) will be quantified.
Time Frame: Up to 48 weeks from the date of randomization
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
percentage of saturation
  Baseline Pre-Dialysis TSAT | 28.1 (8.13) | 27.1 (7.79)
  EoT Pre-Dialysis TSAT | 27.3 (8.52) | 24.0 (7.44)
  Pre-Dialysis TSAT: Change from Baseline to EoT | -1.1 (9.16) | -3.0 (7.70)

13. Secondary Outcome: Variability of Hemoglobin Concentration: Temporal Trend
Description: The mean temporal trend of hemoglobin concentration value changes, as measured weekly from baseline until the end of participation in Stage 2.
Time Frame: Hgb measured weekly; up to 48 weeks from the date of randomization
Population: modified intent to treat: all randomized subjects who received at least one dose of study medication and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: grams per liter per week
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
grams per liter per week | 0.060 (0.298) | 0.002 (0.235)

14. Secondary Outcome: Variability of Hemoglobin Concentration: Residual Standard Deviation
Description: The mean residual standard deviation of hemoglobin concentration value changes, as measured weekly from baseline until the end of participation in Stage 2.
Time Frame: Hgb measured weekly; up to 48 weeks from the date of randomization
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
grams per liter | 4.104 (2.220) | 4.588 (1.949)

15. Primary Outcome: Change From Baseline Hemoglobin at End-of-Treatment: Mean Baseline and End-of-Treatment Hgb
Description: Mean change from baseline Hgb (the average of the three most recent Hgb values preceding randomization) assessments during the last one-sixth of the treatment period for patients who prematurely withdraw from study treatment, but will include a minimum of at least the last two Hgb values. Values expressed are mean baseline and end-of-treatment Hgb, along with the mean difference (standard deviation).
Time Frame: Hgb measured weekly; up to 48 weeks from the date of randomization
Population: modified intent-to-treat: all randomized patients who received at least one dose of study drug and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 148 | 151
grams per liter
  mean baseline hemoglobin | 109.6 (5.91) | 109.0 (6.36)
  mean end-of-treatment hemoglobin | 109.1 (12.53) | 105.2 (13.65)
  mean change in Hemoglobin at end-of-treatment | -0.4 (11.67) | -3.9 (12.52)

ADVERSE EVENTS:
Time Frame: In Stage 2, subjects were randomized to placebo or SFP. They were in Stage 2 for up to 48 weeks. Upon completion of Stage 2, subjects could enter the open-label Stage 3 (all received SFP). The maximum total time on study (Stage 2 + Stage 3) was 72 weeks.
Description: The number of subjects included in the safety population = 300, which is 5 patients fewer than the number of patients randomized. This discrepancy is due to the fact that the Safety population includes only those subjects exposed to study drug. Five subjects withdrew from Stage 2 and 2 subjects withdrew from Stage 3 prior to exposure.
Groups:
- Stage 2 Placebo (Standard Dialysate): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week in Stage 2 for up to 48 weeks.
- Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week in Stage 2 for up to 48 weeks.
- Stage 3 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Upon completion of Stage 2, patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week in Stage 3 for up to 72 weeks of total study participation (Stage 2 + Stage 3).
Arm/Group | Stage 2 Placebo (Standard Dialysate) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 3 Soluble Ferric Pyrophosphate (SFP) in Dialysate
Serious Adverse Events (participants affected / at risk) | 45/151 | 36/149 | 81/205
Other Adverse Events (participants affected / at risk) | 100/151 | 96/149 | 148/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2 Placebo (Standard Dialysate) (N=151) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=149) | Stage 3 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=205)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 0 (0) | 1 (1)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (3)
ARTERIOVENOUS FISTULA ANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA OCCLUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA SITE HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 4 (4)
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
ATRIAL FLUTTER (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 2 (2) | 5 (5)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 5 (8) | 1 (2) | 4 (8)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
CARDIOVERSION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
CATHETER SITE HAEMATOMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 2 (2) | 3 (3)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE DISLOCATION (General disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETIC FOOT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 10 (12) | 2 (2) | 5 (5)
GANGRENE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 (7) | 0 (0) | 9 (11)
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 5 (5)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1) | 4 (4)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
INFECTED SKIN ULCER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 5 (5) | 1 (1) | 3 (3)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
OVARIAN LOW MALIGNANT POTENTIAL TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
PNEUMONIA (Infections and infestations) | 5 (5) | 4 (4) | 5 (10)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
PORTAL HYPERTENSIVE GASTROPATHY (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
RENAL CYST HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL CYST INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
SHOCK (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
STENT-GRAFT ENDOLEAK (General disorders) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VASCULAR GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 4 (6)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2 Placebo (Standard Dialysate) (N=151) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=149) | Stage 3 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=205)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 (6) | 3 (3) | 7 (7)
ANAEMIA (Blood and lymphatic system disorders) | 7 (10) | 3 (4) | 11 (11)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 2 (2) | 7 (7)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 19 (23) | 17 (30) | 25 (58)
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 (3) | 4 (8) | 7 (14)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 7 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (9) | 15 (17)
ASTHENIA (General disorders) | 7 (7) | 7 (7) | 9 (9)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6) | 13 (16)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1) | 11 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 11 (14) | 21 (27)
DECREASED APPETITE (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 8 (8)
DIARRHOEA (Gastrointestinal disorders) | 15 (17) | 13 (14) | 30 (45)
DIZZINESS (Nervous system disorders) | 14 (16) | 13 (17) | 26 (52)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 6 (8) | 22 (34)
FATIGUE (General disorders) | 2 (2) | 7 (7) | 2 (2)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 2 (5) | 5 (7) | 8 (15)
HAEMODIALYSIS-INDUCED SYMPTOM (Injury, poisoning and procedural complications) | 5 (9) | 7 (11) | 39 (199)
HEADACHE (Nervous system disorders) | 8 (9) | 14 (16) | 38 (53)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 4 (6) | 7 (7)
HYPERTENSION (Vascular disorders) | 2 (2) | 3 (3) | 8 (9)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 5 (7) | 5 (5)
INSOMNIA (Psychiatric disorders) | 3 (3) | 0 (0) | 7 (7)
MALAISE (General disorders) | 1 (1) | 2 (2) | 9 (10)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 (20) | 7 (15) | 10 (33)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4) | 13 (16)
NASOPHARYNGITIS (Infections and infestations) | 6 (9) | 2 (2) | 9 (9)
NAUSEA (Gastrointestinal disorders) | 14 (25) | 11 (13) | 20 (31)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 9 (9)
OEDEMA PERIPHERAL (General disorders) | 6 (7) | 8 (12) | 14 (27)
PAIN (General disorders) | 4 (4) | 2 (2) | 10 (11)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (18) | 13 (13)
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1 (2) | 1 (4) | 7 (9)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 41 (216) | 43 (174) | 68 (494)
PYREXIA (General disorders) | 4 (4) | 7 (12) | 10 (11)
THROMBOSIS IN DEVICE (General disorders) | 5 (6) | 3 (3) | 6 (15)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (6) | 4 (4) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 7 (8) | 3 (5)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 4 (8) | 13 (25)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 9 (34)
VOMITING (Gastrointestinal disorders) | 12 (16) | 5 (6) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less